CLINICAL TRIAL: NCT03539211
Title: Clinical Assessment and Thickness Changes of the Oblique and Multifidus Muscles Using a Novel Screening Tool and Exercise Program: A Randomized Controlled Trial
Brief Title: Clinical Assessment and Thickness Changes of the Oblique and Multifidus Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Brian Catania, Physical Therapy Program Manager, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: DDD# 602910
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Abdominal Muscles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotation Exercises (Experimental): 8 minute program of rotation based exercises
  Interventions: Other: Rotation Exercises
- Control Exercises (Active Comparator): 8 minute program of traditional exercises
  Interventions: Other: Control Exercises

INTERVENTIONS:
Other: Rotation Exercises — The subjects received 7 trunk rotation stability exercises x 10 reps each
  Other Names: Sling Activation Session
  Arms: Rotation Exercises
Other: Control Exercises — The subjects received 7 traditional exercises x 10 reps each
  Other Names: Traditional
  Arms: Control Exercises

SUMMARY:
This study evaluates the effect of a rotation based exercise program on core muscle thickness. Additionally, a second aim is to demonstrate the ability of a clinical assessment tool to identify muscle thickness changes. Half of participants receive the rotation based exercises, while the other half perform a traditional core exercise program. It was hypothesized that the rotation based exercises would result in greater changes in muscle thickness.

DETAILED DESCRIPTION:
A number of exercise programs and assessment tools have been evaluated for their ability to influence and measure the core muscles. Inefficient stability and asymmetrical muscle activity of the core have been linked to a wide range of lower extremity injuries. Training of the abdominal muscles to obtain symmetrical recruitment for optimal trunk stabilization is a widespread clinical practice, however valid and reliable assessment tools and effective intervention protocols are lacking. This study uniquely uses both a clinical assessment tool and musculoskeletal ultrasound to measure changes in the core muscles following an exercise intervention. The overall purpose of this study was to design a valid and reliable assessment tool and an effective training protocol to activate the core muscles.

ELIGIBILITY:
Inclusion Criteria:

° Undergraduate and graduate subjects from the University of the Delaware student community.

Exclusion Criteria:

* You could be excluded if you have recently undergone surgery in the last 6 months.
* Currently suffering from low back pain.
* Or have a history of a neurological condition.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea DiTrani, PhD, ATC, Study Director — Neumann University
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotation Exercises | Control Exercises
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotation Exercises | Control Exercises | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (1.5) | 20.7 (1.5) | 20.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Changes in Muscle Thickness
Description: Musculoskeletal ultrasound measured changes in muscle thickness
Time Frame: Baseline and 10 minutes post intervention
Population: External Oblique
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Rotation Exercises | Control Exercises
Number analyzed (Participants) | 16 | 15
centimeters | .820 [.78 to .85] | .671 [.6 to .7]

2. Secondary Outcome: Changes in Clinical Muscle Assessment Using the Novel Sling Screen
Description: Clinician based assessment of muscle function using the sling screen tool; Kappa coefficients were calculated to examine agreement between the 2 physical therapists that completed the sling screen assessments and to account for chance effects in scoring.
  A rating system was used for scoring performance. Min value on the scale is 2 and max value = 5; higher score is a better outcome.
Time Frame: Baseline and 10 minutes post intervention
Population: Anterior Sling
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rotation Exercises | Control Exercises
Number analyzed (Participants) | 16 | 15
score on a scale | -2.02 (.04) | -1.82 (.07)

ADVERSE EVENTS:
Arm/Group | Rotation Exercises | Control Exercises
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes